CLINICAL TRIAL: NCT06846294
Title: OBesity PREVention in Children and Young People Treated with ALLtogetheR: Prehabilitation Feasibility Intervention
Brief Title: Obesity Prevention in Children and Young People Treated for Acute Lymphoblastic Leukaemia with ALLTogether
Acronym: BREVARY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Principal Investigator, Raquel Revuelta Iniesta, Senior Lecturer in Nutrition, University of Exeter
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BREVARY_Mad_Exe
Record Dates: First submitted 2025-01-20; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Diet Intervention; Physical Activity Intervention; Standard Care Control
Keywords: Diet; Physical Activity; Obesity; Acute Lymphoblastic Leukaemia; Children and Young People; ALLTogether
MeSH Terms: conditions — Motor Activity; Obesity; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Diet; Exercise

STUDY DESIGN:
Intervention Model Description: Intervention: online or in hospital Diet: weekly one-to-one sessions for 4 weeks, then fortnightly (8 sessions total). Menus follow Eatwell guide/Food and Agriculture Organization with 20% energy deficit for overweight/obese and equicaloric for healthy weight.
  Physical activity: one-to-one supervised sessions with two-three supervised non-consecutive sessions as tolerated and prescribed based on individual assessment.
  Standard care: diet and physical activity information. Two counselling sessions (psychology) for motivation and adherence.
Masking Description: It is not possible to mask the intervention - as it is diet and physical activity, diet alone or standard care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Diet (Experimental): Individualised Dietary Intervention
  Interventions: Behavioral: Diet
- Diet and Physical Activity (Experimental): Individualised Dietary and Physical Activity Intervention
  Interventions: Behavioral: Diet and physical activity
- Standard Care (No Intervention): No intervention - this is standard care

INTERVENTIONS:
Behavioral: Diet — Individualised dietary intervention
  Arms: Diet
Behavioral: Diet and physical activity — Obesity prevention: Diet, Diet and physical activity and standard care
  Arms: Diet and Physical Activity

SUMMARY:
Background Leukaemia is the most common cancer in children with 800 diagnoses per year in England. To survive, children need strong treatments like chemotherapy and steroids given usually through clinical trials. The current trial used by the NHS is called ALLTogether. Fifty percent of children become obese during treatment due to increased hunger, cravings for junk foods and lack of physical activity. Obesity raises the chance of cancer relapse by 31%, makes treatment side-effects worse and makes it harder to kill off leukaemia cells, which affects how well children do during treatment, as indicated by minimal residual disease, a key predictor of prognosis.

Aims and Objectives This study (called BREVARY) aims to see if we can successfully provide personalised diet and physical activity with behaviour support for children and young people with leukaemia who are being treated with the ALLTogether trial. It will help us figure out if we can perform a bigger study, if this programme could reduce obesity and side-effects and improve survival and wellbeing.

How it will be done We plan to randomly assign participants to one of three groups; one group will get both a diet and physical activity plan, another will get only a diet plan, and the last group will receive standard care. This will take place in Hospital Infantil Universitario Nino Jesus, Madrid and Bristol Royal Hospital for Children and Southwest England NHS-sites. The diet and exercise plans will be created in partnership with the children and their families and delivered online or during regular hospital visits. The diet will follow healthy eating guidelines, consider personal food preferences (including cultural and religious needs), treatment side-effects and personal finances. Assessments of fitness and strength will be taken to plan personalised activities. During the study, the following data will also be collected: weight, height, body fat, diet, biomarkers, microbiome, muscle strength and wellbeing at three different times. "One to one" interviews will be conducted at the end to obtain feedback on their experiences with BREVARY.

This study aims to find out if children and their families/carers are willing to participate in BREVARY, if enough people sign up and stay until the end and if our interventions and health measurements are appropriate.

Potential Impact The results will help determine if a larger study can be performed, if changes are needed and what the cost will be. The study will be disseminated through networks, targeting underserved communities, healthcare professionals and affected families using accessible platforms to spread the word.

DETAILED DESCRIPTION:
The international randomised controlled trial registry shows that no lifestyle intervention (diet, physical activity with integrated counselling) has been performed in the UK. The IDEAL trial performed in the USA demonstrated that diet with energy intake restriction and physical activity was feasible and significantly improved Minimal Residual Disease (MRD) in children diagnosed with Acute lymphoblastic leukaemia (CYP_ALL) and treated with National Cancer Institute/Rome high-risk B-ALL protocol during induction. ALLTogether is similar and will for the first time provide an excellent platform to prevent obesity in CYP_ALL.

Obesity associated relapse is attributed to adipocyte-mediated chemo-resistance, which occurs in CYP_ALL with higher fat mass and leads to more persistent MRD. MRD is a marker of leukaemic cells and the strongest predictor of prognosis including both remission and relapse. Therefore, obesity is identified as a prognostic factor for relapse (measured by MRD) and it is associated with increased morbidity and mortality, and poorer wellbeing.

Only two dietary feasibility interventions have investigated CYP_ALL differing in the type (diet alone vs. diet and physical activity) and the length of intervention (1 - 6 months). Both showed improvements in diet quality, high participation (>70%) and 56 - 82% adherence. Indeed, the IDEAL trial also showed improvements in MRD and body composition, making it suitable to base BREVARY's design. Consensus exists regarding using patient-centre interventions in clinical settings; like the Individualised Macronutrient Meal-Equivalent Menu (Menus). This approach reduces food associated stress, anxiety and financial costs, while empowering patients and their families/carers, thus improving adherence. It has been shown to be successful in adults with breast cancer and provides a validated approach to CYP_ALL.

A systematic review showed that individualised physical activity combining fitness and strength mitigated complications in CYP_ALL. However, it was difficult to draw firm conclusions because evidence were limited by sample sizes, adherence was seldom reported and study designs were heterogenous differing in length (1 - 30 months), exercise type and intensity and assessed outcomes (e.g. cardiorespiratory fitness, strength and wellbeing). Six trials are underway including all cancers with interventions being either individualised ("as able" and play-based exercise for children aged <5 years) or employing generic exercise prescriptions with intensity "as able". They are investigating fitness, strength and wellbeing; however, none have incorporated dietary assessment or intervention.

4. Research proposal

Aim

Investigate the feasibility of conducting a randomised controlled trial (RCT) to prevent obesity in CYP_ALL and treated with ALLTogether.

The hypothesis is that BREVARY will reduce obesity rates, improve clinical outcomes by reducing side-effects and relapse and improving CYP_ALL and their families/carers' quality of life. BREVARY will establish if a multi-site RCT is feasible and acceptable to families and clinical teams, examine recruitment and data collection strategies, and assess candidate outcomes.

BREVARY comprises three workstreams (WS):

WS1: Implementing a RCT of BREVARY for 3 months involving newly diagnosed CYP_ALL treated with ALLTogether in SW England NHS-sites and Hospital Infantil Universitario Nino Jesus Madrid WS2: Process evaluation of BREVARY RCT examining feasibility and maintenance of intervention (3 months intervention, maintenance at 6 months) WS3: Assessment of feasibility of progression to a definitive trial, including setting trial parameters

Objectives

* Assess recruitment, including acceptability of randomisation to stakeholders, across ethnically, geographically and socially diverse communities (WS1)
* Assess interventions acceptability and retention (WS1/WS2)
* Assess feasibility and appropriateness of quantitative and qualitative outcomes (WS1)
* Assess RCT resource implications of interventions and potential service use savings (WS1/WS3)
* Assess fidelity and adherence to protocol within interventions and control groups (WS1/WS2)
* Assess feasibility of progression to a definitive trial, set out main parameters and estimate both sample size and cost of a RCT (WS3)

Project plan

WS1: Implementing BREVARY

Study design BREVARY is phase 2 of Medical Research Council framework for complex interventions. Development and identification of the complex intervention (phase 1) was performed based on the IDEAL pilot-trial. BREVARY was designed in consultation with NIHR Nutrition and Cancer and PPI, reviewed by NIHR RSS and is supported by ALLTogether sponsors (UK and Spain).

Feasibility three-arm non-blinded parallel RCT with integrated quantitative and qualitative measures. Quantitative measures will be performed at baseline, end of induction (4 - 6 weeks) and during consolidation treatment (3 months weeks) and a follow up at 6 months. Qualitative measures will be performed at the end of BREVARY in a sample subgroup. The three-arms include combined diet and physical activity, diet only and standard care.

Recruitment Recruitment will be conducted by researchers. Inclusion criteria

* CYP aged between 2 - 21 years.
* Newly diagnosed and relapse CYP_ALL treated in University Hospital Bristol and Weston NHS Foundation Trust and Hospital Infantil Universitario Nino Jesus, Madrid
* Within two weeks of being recruited to ALLTogether.
* Treated with curative intent. Exclusion criteria
* CYP not partaking in ALLTogether.
* CYP treated with palliative intent.
* Those excluded by NHS-staff for clinical reasons. BREVARY aims to recruit 10 - 15 in each arm and each international centre (n= 60 - 90 in SW England and Madrid; 50% recruitment rate, which is below previous studies and the IDEAL trial to test feasibility and to calculate the variability of reliable estimates of continuous variables.

Eligible participants will be randomised using computer-generated restricted (nutritional status, age and sex) randomisation procedure in 1:1:1 ratio.

BREVARY Intervention (table 1)

Twenty % energy deficit and equicaloric intervention will be applied to those classified as overweight/obese and healthy weight respectively by diet (- 20%).

Researchers will deliver weekly one-to-one supervised sessions during induction and fortnightly during consolidation (total 8 sessions) online/home or at routine appointments. Physical activity intervention will include two additional sessions supervised non-consecutive sessions as tolerated. Both designed following PPI preferences.

Dietary intervention Menus based on Eatwell guide in the UK and Food and Agriculture Organisation in Spain will be used. Menus consists of prescribing 7 interchangeable meal options matched in energy and macronutrients requirements to reduce participants meal planning burden. It accounts for side-effects, psycho-social factors and religious, cultural, personal (and PPI) preferences. Nutritics® will be used to create Menus and estimate nutrients.

CYP_ALL referred to Dietetics will receive the intervention post-Dietetic discharged to avoid interference with nutritional support.

Physical activity intervention Individualised plans will be prescribed based on fitness and clinical condition. The programme will start at enrolment unless contraindicated. Sessions will include a combination of aerobic, balance and resistance exercise based on individual fitness and strength, age and clinical history as well as individual preferences and available equipment.

Standard care CYP_ALL will receive usual care (described in "The problem"). Counselling sessions for CYP_ALL and families/carers (all groups) Counselling sessions were requested by PPI and are recommended for motivation and adherence in long-term clinical interventions.

Two online/home (or at routine appointments) one-to-one sessions will be delivered. Sessions will be designed by all co-applicants, reviewed by our clinical psychologist and delivered by the researchers with PPI CoA support and focusing on:

(i) Diet and physical activity benefits (ii) Behaviour and autonomy (iii) Difficulties encountered and how to address them (iv) Motivation Data collection (all groups)

* Eligible CYP_ALL
* Eligible CYP_ALL approached to participate
* Families declining intervention before randomisation, after randomisation and after the first set of measurements (before follow-ups)
* Families allocated to interventions dropping out between second and final follow-up
* Families allocated to standard care dropping out between second and final follow-up

Health Electronic Records (HER) will be accessed to collect demographics (CYP_ALL sex, ethnicity and age), socio-economics (parents' relationship status, siblings, employment status, education level, income and housing status), clinical (diagnosis, treatments, side-effects, hospital admissions), routine biomarkers (MRD, immunoglobulins, full blood count, total cholesterol, high density lipoprotein and low density lipoprotein and glucose) and other biomarkers (leptin and adiponectin) and stool samples (microbiome). Participants' postcodes will be linked to the Indices of Multiple Deprivation.

Based on the IDEAL trial, feasibility and acceptability and PPI feedback, the following outcome measures will be taken at baseline, 4 - 6 weeks, 3 months and a follow up at 6 months (to assess intervention sustainability - no intervention from 3 - 6 months).

* Weight, height and body composition (Multi-frequency Bio-electrical Impedance)
* Dietary intake using a multiple-pass 24 hour recall
* Seven days physical activity levels at each follow up using GENEActiv accelerometers, strength by hand-held hydraulic dynamometer and fitness by 15-foot walk (excluding children aged <5y).
* CYP_ALL and their families/carers' QoL will be assessed at baseline and at completion using two validated questionnaires PedQL-Cancer and Parents PedQL-Cancer.

We will determine primary and secondary candidate outcome measures for future trial based on performance of selected measures.

Candidate primary outcome measures for definitive trial

* Body mass index Z-score (≤ 19 years)
* Muscle and fat mass percentage
* MRD
* Quality of Life: PedQL-Cancer and Parents PedQL-Cancer Candidate secondary outcome measures for definitive trial
* Biomarkers and Microbiome
* Food group indicators and nutrient intake
* Physical activity levels
* Hand strength (percentiles 5 ≤ 18 years)
* CPET - Fitness excluding children aged < 5 years
* Clinical outcomes, number and type of treatment side-effects and intervention side-effects
* Hospital admissions
* Changes in treatment regime (ALLTogether)
* Microbiome: composition and diversity of microbiome

Analysis CONSORT flow diagram will be used to report participant flow and descriptive statistics for demographics, clinical and socio-economic data with overall data and stratified by arm. Appropriate distribution or frequencies will be used (count/percentages, mean/SD and median/IQR). IBM_SPSS statistics® will be used for analysis and a Statistical Analysis Plan will be signed-off prior to any analysis taking place.

WS2: Process evaluation The process evaluation assesses how implementation of BREVARY is achieved, influenced by contextual factors including randomisation and trial design, and quality of implementation and acceptability. The following stakeholders will be included: Parents/carers whose CYP_ALL partake in BREVARY, CYP_ALL able to understand the questions and communicate an answer and researchers plus NHS-staff directly involved in implementing BREVARY. RE-AIM (http://www.re-aim.org/) based on reach, effectiveness, adoption, implementation and maintenance will be used.

Semi-structured one-to-one online (or at routine appointment) interviews will be conducted to a subgroup (n = 15) with equal representation from each arm to explore enjoyment:

* Best and worst things about partaking
* Overall satisfaction
* Likelihood to recommend BREVARY
* Reasons for dropping out Facilitator records will be completed by the researchers using structured case-records to collect RE-AIM

Analysis Quantitative survey data will be analysed using descriptive statistics. Free text responses will be analysed using thematic analysis and audio recordings will be transcribed, anonymised and data analysed using thematic analysis in Nvivo®.

Fidelity: Intervention delivery (usage statistics), receipt (usage statistics and interviews) and enactment (interviews, questionnaires and measurements) as well as repeated engagement (usage statistics and counselling sessions) will be conducted separately. Findings will be integrated following a triangulation protocol to assess whether data agree (convergence), complement one another (complementary), or contradict each other (dissonance).

WS3: Progression criteria and definitive RCT design

Results from WS1 and WS2 will be reviewed by all co-applicants. A trial will be regarded feasible if the following criteria are met:

Progression criteria and definitive RCT design

* Recruitment rate ≥ 50%
* ≥ 70% of recruited families complete the trial in one of the intervention groups
* ≥ 70% of families, researchers and clinical staff agree that the intervention is acceptable (RE-AIM)
* Recruited participants complete ≥ 60% of the supervised sessions (RE-AIM)
* ≥ 70% of families agree that the intervention is enjoyable

Health economics Within-trial economic and resource use analysis based on complex intervention protocols will be used. This reduces participants' burden and meets PPI feedback.

The within-trial analysis will investigate the cost-effectiveness of each arm. The primary within-trial analysis used in the full trial will be a cost-utility-analysis (CUA), which estimates the incremental cost per quality adjusted life (QALY) of each arm. QALY will be generated via measurement of utility values using PedsQL-cancer and Parents PedQL-Cancer instrument mapped to the EQ-5D.

The resource use analysis will be estimated using HER. Data (e.g. admissions, medication) will be collected by researchers. A cost-consequences framework will be used to describe resources used and benefits gained from the intervention without developing a full cost-effectiveness estimate.

ELIGIBILITY:
Inclusion Criteria:

* CYP aged between 5 - 21 years.
* Newly diagnosed or relapsed CYP_ALL treated in University Hospital Bristol and Weston NHS Foundation Trust and Hospital Infantil Universitario Nino Jesus, Madrid
* Within two weeks of being recruited to ALLTogether.
* Treated with curative intent.

Exclusion Criteria:

* CYP not partaking in ALLTogether.
* CYP treated with palliative intent.
* Those excluded by healthcare professionals or clinical reasons

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Minimal Residual Disease | initial assessment, day 29, day 50 and day 78
  Candidate Primary Outcome (feasibility study). Hospital own's laboratory assay
Muscle and fat mass | Initial assessment, at 29 days, at 3 months, at 6 months
  Candidate primary outcome, Multifrequency BIA FFM and FM percentage Impedance Reactant
Body Mass Index Z score | initial assessment, at day 29, at 3 months and at 6 months
  Candidate Primary Outcome Calculated from weight and height (weight/height^2) WHO BMI Z score (scale score) Z-Score Range Nutritional Status < -3 SD: Severe undernutrition (Severely underweight, stunted, or wasted)
  * -3 SD and < -2 SD: Moderate undernutrition (Underweight, stunted, or wasted)
  * -2 SD and ≤ +1 SD: Healthy weight (Normal nutritional status)
    * +1 SD and ≤ +2 SD: Overweight
    * +2 SD: Obese
Quality of Life | initial assessment, at 3 months and at 6 months
  Candidate Primary outcome (Quality of Life: PedQL-Cancer Module questionnaire) The PedsQL-Cancer Module includes multiple subscales that address specific areas of functioning and challenges related to cancer, such as: Pain and hurt, Nausea, Procedural anxiety, Treatment anxiety, Worry, Cognitive problems, Perceived physical appearance, Communication.
  To calculate scores, the items are reverse scored and linearly transformed to a Original Response Reverse Score (Transformed Score) 0 = Never 100
  1. = Almost Never 75
  2. = Sometimes 50
  3. = Often 25
  4. = Almost Always 0
  Scores are reverse, thus higher scores indicate better health-related quality of life or fewer reported problems.
  Mean scores are calculated for each subscale by summing the item scores and dividing by the number of items answered. If more than 50% of the items in a subscale are missing, the subscale score is not computed.
Parent's quality of life | Initial assessment, at 3 months and at 6 months
  Parents PedQL-Cancer he PedsQL Cancer Module - Parent Proxy Report is a specialized tool designed to assess health-related quality of life (HRQoL) in children and adolescents with cancer, based on the parent's perception.
  The Parent PedsQL Cancer Module includes the following subscales tailored to cancer-related challenges: Pain and Hurt, Nausea, Procedural Anxiety, Treatment Anxiety, Worry, Cognitive Problems, Perceived Physical Appearance, Communication To calculate scores, the items are reverse scored and linearly transformed to a 0-100 scale: 0 = 100; 1 = 75; 2 = 50; 3 = 25; 4 = 0 Higher scores indicate better health-related quality of life or fewer reported problems.
Feasibility: Participation rate | Baseline, time 0
  The proportion of the target population that actually participates in the intervention measured in frequencies
Feasibility: Representativeness | At 0, day 29, 3 months and 6 months
  The degree to which the participants reflect the broader population intended to benefit from the intervention.
  Outcome measure in percentages
Feasibility: Accessibility | At 0, day 29, 3 months and 6 months
  Evaluates whether the intervention is accessible to all segments of the target population, including those who are typically underrepresented.
  Outcome measure in percentage
Feasibility: Barriers to participation | At 0, day 29, 3 months and 6 months
  Identifies factors that prevent individuals from engaging with the intervention, such as lack of awareness, logistical issues, or cultural barriers.
  Outcome: qualitative
Feasibility: Effectiveness | At 0, day 29, 3 months and 6 months
  The trial will be regarded feasible if the following criteria are met:
  * Recruitment rate ≥ 50%
  * ≥ 70% of recruited families complete the trial in one of the intervention groups
  * ≥ 70% of families, researchers and clinical staff agree that the intervention is acceptable (survey)
  * Recruited participants complete ≥ 60% of the supervised sessions
  * ≥ 70% of families agree that the intervention is enjoyable The overall outcome is categorical: Yes, No or yes with conditions/amendments
Feasibility: Adoption | At 0, day 29, 3 months and 6 months
  Settings: the proportion of settings that agree to implement the intervention. Outcome measured in percentage.
Feasibility: staff/provider adoption | At 0, day 29, 3 months and 6 months
  The proportion and characteristics of researchers and healthcare staff who choose to deliver the intervention.
  Outcome in percentages
Feasibility: Barriers and facilitators: Qualitative | At 0, day 29, 3 months and 6 months
  Identifies factors that help or hinder the willingness of organisations and individuals to adopt the intervention (e.g., cost, training requirements, organisational culture).
  Outcome: quaitative
Feasibility: Fidelity | At 0, day 29, 3 months and 6 months
  Fidelity scores ranging from 0 to 100 (e.g., percentage of protocol elements followed) where 0 is nothing was followed and 100 everything was followed as originally planned.
Cost-effectiveness | At 0, 3 months and 6 months
  Cost-utility analysis to evaluate the economic value of different interventions (or arms) by comparing their costs to their outcomes. This is based on quality-adjusted life in years. QALY will be generated via measurement of utility values using PedsQL-cancer and Parents PedQL-Cancer instrument mapped to the EQ-5D.
  Outcome: scale in pounds and euros. Total cost of control, cost of diet alone and cost of diet and physical activity

SECONDARY OUTCOMES:
Leptin | Initial assessment, at day 29, at 3 months and at 6 months
  Candidate secondary outcomes for future RCT: leptin (abcam assay)
Food group indicators and nutrient intake | Initial assessment, at day 29, at 3 months and at 6 months
  Candidate Secondary Outcome for RCT multiple pass 24-hour recall Food groups (Eatwell Guide and A healthy eating index score (HEI)) Macronutrients and micronutrients (analysed in Nutritics) compared to UK Dietary Recommended Daily Intake (DRVs 1991, SANC 2011) and Spanish Ingestas Nutricionales de Referencia (AESAN 2019)
Physical activity levels min/day | Initial assessment, at 3 months and at 6 months
  Candidate secondary outcome for RCT GENEActiv accelerometers (min/day) 5 week days, 2 weekend days (minimum recorded 10 hours)
Handgrip strength | Initial assessment, at day 29, at 3 months and at 6 months
  Candidate secondary outcome for RCT hand-held hydraulic dynamometer
Fitness | Initial assessment, at day 29, at 3 months and at 6 months
  15-foot walk
Side-effects | Throughout the study (0 - 3 months), then again at 6 months
  Candidate Secondary Outcome for RCT: treatment side-effects, intervention arms side-effects, hospital admissions (and length), changes in treatment regime (ALLTogether)
Gut microbiome composition | Initial assessment and 3 months
  Characterisation of gut microbiome composition: α- and β-diversity, relative abundances (comparison between groups) 16sRNA sequencing
Adiponectin | Initial assessment, at day 29, at 3 months and at 6 months
  Candidate secondary outcome for RCT, Abcam assay
Insulin | Initial assessment, at day 29, at 3 months and at 6 months
  Candidate secondary outcome for RCT, Oxford Biosyste ELISA
Immunoglobulin A (IgA) | Initial assessment, at day 29, at 3 months and at 6 months
  IgA (hospital owns assays)
Immunoglobulin G (IgG) | Initial assessment, at day 29, at 3 months and at 6 months
  IgG - hospital own's laboratory
Immunoglobulin M (IgM) | Initial assessment, at day 29, at 3 months and at 6 months
  IgM (hospital own's assay)
Total Cholesterol | Initial assessment, at day 29, at 3 months and at 6 months
  Total Cholesterol (TCh) - hospital owns assay
High Density Lipoprotein (HDL) | Initial assessment, at day 29, at 3 months and at 6 months
  HDL (hospital own's assay)
Low Density Lipoprotein (LDL) | Initial assessment, at day 29, at 3 months and at 6 months
  LDL (hospital's own assay)
Triglycerides (TGA) | Initial assessment, at day 29, at 3 months and at 6 months
  TGA (hospital's own assay)
Glucose | Initial assessment, at day 29, at 3 months and at 6 months
  Glucose (hospital's own assay)
C-Reactive Protein (CRP) | Initial assessment, at day 29, at 3 months and at 6 months
  Standard Sensitivity CRP, hospital's own assay.

OTHER OUTCOMES:
Characterisation of gut microbiome: Diversity | At 0, day 29, 3 months and 6 months
  Outcome from 16sRNA sequencing: alpha and beta bacteria.
Gut microbiome: Relative abundance | At 0, day 29, 3 months and 6 months
  Relative abundances (comparison between groups: alpha and beta bacteria)

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Revuelta Iniesta, PhD, Study Chair — University of Exeter; Carmen Fiuza Luces, PhD, Study Chair — Hospital 12 de Octubre Research Institute; Raquel Revuelta Iniesta, PhD, Study Director — University of Exeter
Locations (2):
- Hospital Infantil Universitario Nino Jesus, Madrid, Madrid, Spain
- University Hospitals Bristol & Weston NHS Trust, Bristol, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Given the sensitive nature of hospital patient data and the feasibility focus of your study, sharing individual participant data does not align with ethical guidelines, data protection regulations, and the consent provided by participants.

REFERENCES:
- [Background] Khan KA, Petrou S, Rivero-Arias O, Walters SJ, Boyle SE. Mapping EQ-5D utility scores from the PedsQL generic core scales. Pharmacoeconomics. 2014 Jul;32(7):693-706. doi: 10.1007/s40273-014-0153-y. PMID 24715604
- [Background] O'Cathain A, Murphy E, Nicholl J. Three techniques for integrating data in mixed methods studies. BMJ. 2010 Sep 17;341:c4587. doi: 10.1136/bmj.c4587. No abstract available. PMID 20851841
- [Background] Arnetz J, Sudan S, Goetz C, Arnetz B, Gowland L, Manji S, Ghosh S. Preliminary development of a questionnaire measuring patient views of participation in clinical trials. BMC Res Notes. 2019 Oct 21;12(1):667. doi: 10.1186/s13104-019-4724-z. PMID 31639069
- [Background] Deidda M, Boyd KA, Minnis H, Donaldson J, Brown K, Boyer NRS, McIntosh E; BeST study team. Protocol for the economic evaluation of a complex intervention to improve the mental health of maltreated infants and children in foster care in the UK (The BeST? services trial). BMJ Open. 2018 Mar 14;8(3):e020066. doi: 10.1136/bmjopen-2017-020066. PMID 29540420
- [Background] Braun V, Clarke V (2006) Using thematic analysis in psychology. Qual. Res.Psychol 3, 77-101
- [Background] Fielding D, Duff A. Compliance with treatment protocols: interventions for children with chronic illness. Arch Dis Child. 1999 Feb;80(2):196-200. doi: 10.1136/adc.80.2.196. No abstract available. PMID 10325743
- [Background] Gibson AA, Sainsbury A. Strategies to Improve Adherence to Dietary Weight Loss Interventions in Research and Real-World Settings. Behav Sci (Basel). 2017 Jul 11;7(3):44. doi: 10.3390/bs7030044. PMID 28696389
- [Background] Varni JW, Katz ER, Seid M, Quiggins DJ, Friedman-Bender A, Castro CM. The Pediatric Cancer Quality of Life Inventory (PCQL). I. Instrument development, descriptive statistics, and cross-informant variance. J Behav Med. 1998 Apr;21(2):179-204. doi: 10.1023/a:1018779908502. PMID 9591169
- [Background] Varni JW, Burwinkle TM, Katz ER, Meeske K, Dickinson P. The PedsQL in pediatric cancer: reliability and validity of the Pediatric Quality of Life Inventory Generic Core Scales, Multidimensional Fatigue Scale, and Cancer Module. Cancer. 2002 Apr 1;94(7):2090-106. doi: 10.1002/cncr.10428. PMID 11932914
- [Background] Rehorst-Kleinlugtenbelt LB, et al. (2019) Physical activity level objectively measured by accelerometery in children undergoing cancer treatment at home and in a hospital setting: A pilot study. J. Pediatr. Hematol. Oncol. 4, 82-88
- [Background] Russell DJ, Rosenbaum PL, Cadman DT, Gowland C, Hardy S, Jarvis S. The gross motor function measure: a means to evaluate the effects of physical therapy. Dev Med Child Neurol. 1989 Jun;31(3):341-52. doi: 10.1111/j.1469-8749.1989.tb04003.x. PMID 2753238
- [Background] Reilly JJ, Montgomery C, Jackson D, MacRitchie J, Armstrong J. Energy intake by multiple pass 24 h recall and total energy expenditure: a comparison in a representative sample of 3-4-year-olds. Br J Nutr. 2001 Nov;86(5):601-5. doi: 10.1079/bjn2001449. PMID 11737958
- [Background] Kang M, Ragan BG, Park JH. Issues in outcomes research: an overview of randomization techniques for clinical trials. J Athl Train. 2008 Apr-Jun;43(2):215-21. doi: 10.4085/1062-6050-43.2.215. PMID 18345348
- [Background] R. RDAHI (2015) Complex Interventions in Health: An Overview of Research Methods. 1st ed. Oxford: Routledge
- [Background] Pasquet M (2022) Adapted Physical Activity for Children Treated With Cancer and Insulin Sensitivity (APACIS).
- [Background] Mochel J (2021) LCI-PED-NOS-EXER-001: Exercise in Pediatric Oncology Patients.
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508
- [Background] Culos-Reed NS (2021) IMPACT: Implementation of Physical Activity for Children.
- [Background] Limon-Miro AT, Lopez-Teros V, Astiazaran-Garcia H. Dynamic Macronutrient Meal-Equivalent Menu Method: Towards Individual Nutrition Intervention Programs. Methods Protoc. 2019 Sep 5;2(3):78. doi: 10.3390/mps2030078. PMID 31491882
- [Background] López Teros V (2021) Nutritional Intervention in Acute Lymphoblastic Leukemia (ALL).
- [Background] Friend AJ, Feltbower RG, Hughes EJ, Dye KP, Glaser AW. Mental health of long-term survivors of childhood and young adult cancer: A systematic review. Int J Cancer. 2018 Sep 15;143(6):1279-1286. doi: 10.1002/ijc.31337. Epub 2018 Mar 15. PMID 29468674
- [Background] Egnell C, Heyman M, Jonsson OG, Raja RA, Niinimaki R, Albertsen BK, Schmiegelow K, Stabell N, Vaitkeviciene G, Lepik K, Harila-Saari A, Ranta S. Obesity as a predictor of treatment-related toxicity in children with acute lymphoblastic leukaemia. Br J Haematol. 2022 Mar;196(5):1239-1247. doi: 10.1111/bjh.17936. Epub 2021 Nov 2. PMID 34726257
- [Background] Borowitz MJ, Devidas M, Hunger SP, Bowman WP, Carroll AJ, Carroll WL, Linda S, Martin PL, Pullen DJ, Viswanatha D, Willman CL, Winick N, Camitta BM; Children's Oncology Group. Clinical significance of minimal residual disease in childhood acute lymphoblastic leukemia and its relationship to other prognostic factors: a Children's Oncology Group study. Blood. 2008 Jun 15;111(12):5477-85. doi: 10.1182/blood-2008-01-132837. Epub 2008 Apr 3. PMID 18388178
- [Background] Walters M, Mowbray C, Jubelirer T, Jacobs S, Kelly KM, Smith K, Yao Y, Jin Z, Ladas EJ. A bilingual dietary intervention early in treatment is feasible and prevents weight gain in childhood acute lymphoblastic leukemia. Pediatr Blood Cancer. 2021 May;68(5):e28910. doi: 10.1002/pbc.28910. Epub 2021 Feb 15. PMID 33590674
- [Background] Limon-Miro AT, Valencia ME, Lopez-Teros V, Aleman-Mateo H, Mendez-Estrada RO, Pacheco-Moreno BI, Astiazaran-Garcia H. An individualized food-based nutrition intervention reduces visceral and total body fat while preserving skeletal muscle mass in breast cancer patients under antineoplastic treatment. Clin Nutr. 2021 Jun;40(6):4394-4403. doi: 10.1016/j.clnu.2021.01.006. Epub 2021 Jan 9. PMID 33485708
- [Background] Belanger V, Delorme J, Napartuk M, Bouchard I, Meloche C, Curnier D, Sultan S, Laverdiere C, Sinnett D, Marcil V. Early Nutritional Intervention to Promote Healthy Eating Habits in Pediatric Oncology: A Feasibility Study. Nutrients. 2022 Feb 28;14(5):1024. doi: 10.3390/nu14051024. PMID 35267999
- [Background] Orgel E, Framson C, Buxton R, Kim J, Li G, Tucci J, Freyer DR, Sun W, Oberley MJ, Dieli-Conwright C, Mittelman SD. Caloric and nutrient restriction to augment chemotherapy efficacy for acute lymphoblastic leukemia: the IDEAL trial. Blood Adv. 2021 Apr 13;5(7):1853-1861. doi: 10.1182/bloodadvances.2020004018. PMID 33792627
- [Background] Braam KI, van der Torre P, Takken T, Veening MA, van Dulmen-den Broeder E, Kaspers GJ. Physical exercise training interventions for children and young adults during and after treatment for childhood cancer. Cochrane Database Syst Rev. 2016 Mar 31;3(3):CD008796. doi: 10.1002/14651858.CD008796.pub3. PMID 27030386
- [Background] Revuelta Iniesta R, Gerasimidis K, Paciarotti I, McKenzie JM, Brougham MF, Wilson DC. Micronutrient status influences clinical outcomes of paediatric cancer patients during treatment: A prospective cohort study. Clin Nutr. 2021 May;40(5):2923-2935. doi: 10.1016/j.clnu.2021.03.020. Epub 2021 Mar 20. PMID 33964502
- [Background] Glatt D, Hughes C, McCarthy O, O'Shea F, Brougham MFH, Wilson DC, Revuelta Iniesta R. Nutritional screening and assessment of paediatric cancer patients: A quality improvement project (baseline results). Clin Nutr ESPEN. 2020 Aug;38:242-252. doi: 10.1016/j.clnesp.2020.04.003. Epub 2020 Apr 27. PMID 32690165
- [Background] Ren Y, Li X. Direct and indirect costs of families with a child with acute lymphoblastic leukaemia in an academic hospital in China: a cross-sectional survey. BMJ Open. 2019 Jul 18;9(7):e030511. doi: 10.1136/bmjopen-2019-030511. PMID 31324687
- [Background] Rahiala J, Riikonen P, Kekalainen L, Perkkio M. Cost analysis of the treatment of acute childhood lymphocytic leukaemia according to Nordic protocols. Acta Paediatr. 2000 Apr;89(4):482-7. doi: 10.1080/080352500750028230. PMID 10830464
- [Background] Soliman R, Heneghan C, Bolous NS, Sidhom I, Ahmed S, Roberts N, Oke J, Elhaddad A. Systematic review of costs and cost-effectiveness of treatment for relapsed/refractory acute leukemia in children and young adults. Expert Rev Hematol. 2022 Apr;15(4):345-357. doi: 10.1080/17474086.2022.2069096. Epub 2022 May 4. PMID 35485262
- [Background] Orgel E, Tucci J, Alhushki W, Malvar J, Sposto R, Fu CH, Freyer DR, Abdel-Azim H, Mittelman SD. Obesity is associated with residual leukemia following induction therapy for childhood B-precursor acute lymphoblastic leukemia. Blood. 2014 Dec 18;124(26):3932-8. doi: 10.1182/blood-2014-08-595389. Epub 2014 Oct 27. PMID 25349177
- [Background] Brinksma A, Sanderman R, Roodbol PF, Sulkers E, Burgerhof JG, de Bont ES, Tissing WJ. Malnutrition is associated with worse health-related quality of life in children with cancer. Support Care Cancer. 2015 Oct;23(10):3043-52. doi: 10.1007/s00520-015-2674-0. Epub 2015 Mar 10. PMID 25752883
- [Background] Lovell AL, Gardiner B, Henry L, Bate JM, Brougham MFH, Iniesta RR. The evolution of nutritional care in children and young people with acute lymphoblastic leukaemia: a narrative review. J Hum Nutr Diet. 2025 Feb;38(1):e13273. doi: 10.1111/jhn.13273. Epub 2024 Jan 7. PMID 38185902
- [Background] Coombs A, Schilperoort H, Sargent B. The effect of exercise and motor interventions on physical activity and motor outcomes during and after medical intervention for children and adolescents with acute lymphoblastic leukemia: A systematic review. Crit Rev Oncol Hematol. 2020 Aug;152:103004. doi: 10.1016/j.critrevonc.2020.103004. Epub 2020 May 27. PMID 32580035
- [Background] Oeffinger KC, Mertens AC, Sklar CA, Yasui Y, Fears T, Stovall M, Vik TA, Inskip PD, Robison LL; Childhood Cancer Survivor Study. Obesity in adult survivors of childhood acute lymphoblastic leukemia: a report from the Childhood Cancer Survivor Study. J Clin Oncol. 2003 Apr 1;21(7):1359-65. doi: 10.1200/JCO.2003.06.131. PMID 12663727
- [Background] Iniesta RR, Paciarotti I, Brougham MF, McKenzie JM, Wilson DC. Effects of pediatric cancer and its treatment on nutritional status: a systematic review. Nutr Rev. 2015 May;73(5):276-95. doi: 10.1093/nutrit/nuu062. Epub 2015 Mar 29. PMID 26011902
- [Background] Revuelta Iniesta R, Paciarotti I, Davidson I, McKenzie JM, Brougham MFH, Wilson DC. Nutritional status of children and adolescents with cancer in Scotland: A prospective cohort study. Clin Nutr ESPEN. 2019 Aug;32:96-106. doi: 10.1016/j.clnesp.2019.04.006. Epub 2019 May 17. PMID 31221298
- [Background] Cohen J, Collins L, Gregerson L, Chandra J, Cohn RJ. Nutritional concerns of survivors of childhood cancer: A "First World" perspective. Pediatr Blood Cancer. 2020 Jun;67 Suppl 3:e28193. doi: 10.1002/pbc.28193. Epub 2020 Jan 29. PMID 31994836
- [Background] Malard F, Mohty M. Acute lymphoblastic leukaemia. Lancet. 2020 Apr 4;395(10230):1146-1162. doi: 10.1016/S0140-6736(19)33018-1. PMID 32247396
- Available data/document: Protocol and ethics can be shared on request — https://medicine.exeter.ac.uk/phss/research/foodnutrition/clinical/ — Information will be shared following ethical approval on relevant websites